CLINICAL TRIAL: NCT00203047
Title: A Multi-Centered, Randomized, Double-Blind, Placebo Controlled Study Assessing the Add-on Effect of Oral Steroids in Relapsing Remitting Multiple Sclerosis Subjects Treated With Glatiramer Acetate (GA)
Brief Title: Assessment Study of Steroid Effect in Relapsing Multiple Sclerosis Subjects Treated With Glatiramer Acetate
Acronym: ASSERT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment decreased sample size; No unexpected safety issues.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNC GA MS 2004_01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; brain atrophy; Glatiramer Acetate; Copaxone; Steroids; Prednisone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Glatiramer Acetate; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GA + Placebo (Active Comparator): Glatiramer acetate (GA) 10mg as a subcutaneous injection daily, plus a placebo to mimic prednisone given daily.
  Interventions: Drug: Glatiramer Acetate; Drug: Placebo
- GA + Prednisone (Experimental): Glatiramer acetate (GA) 20mg daily as a subcutaneous injection, plus 1250 mg of prednisone daily.
  Interventions: Drug: Glatiramer Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Glatiramer Acetate — 20mg glatiramer acetate (GA) administered by daily subcutaneous injections
  Other Names: Copaxone
Drug: Placebo — Placebo for prednisone given daily
  Arms: GA + Placebo
Drug: Prednisone — Prednisone 1250 mg taken daily
  Other Names: corticosteroid
  Arms: GA + Prednisone

SUMMARY:
This is a study evaluating the effect on brain volume of daily glatiramer acetate (GA) and add-on pulse steroids.

DETAILED DESCRIPTION:
One interim analysis was planned for possible early termination due to proven efficacy when 75% of the preplanned 500 (approx. 375 patients) recruited patients completed the entire study duration or early discontinued.

In addition to the stopping rule already given for proven efficacy, the sponsor was also interested in examining the data for futility (i.e., absence of the desired treatment effect) with the view to terminating the trial if an "insufficient" effect of the treatment is seen. The reasons why the need for futility arose were:

1. Recruitment difficulties
2. Increasing dropout rate
3. Budgetary constraints

The primary efficacy measure is defined as the percent change from baseline to termination (Month 36 or Early Termination) in normalized brain volume (Brain Atrophy) measured according to the SIENA (Structural Imaging Evaluation using Normalization of Atrophy) method. However, since not many patients had completed the entire study at the time of futility analysis, it was the sponsor's decision that the futility analysis be performed on patients with MRI scans at months 24 or 36 or at early termination visits - the latest available.

Based on the recalculation of study power (probability is unconditioned on the interim result and provide the real power of the study if designed anew), conditional power (based on the interim results) and risk assessment of a false negative, the Data Monitoring Committee agreed that the study should be terminated early.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite multiple sclerosis (CDMS) according to Poser (Ann. Neurol. 1983) or McDonald (Ann. Neurol. 2001)
2. Subjects eligible for GA treatment based on the investigator's clinical assessment and according to the current indication.
3. Subjects must have a relapsing remitting disease course.
4. Subjects must have had at least 1 documented relapse within the last year prior to study entry.
5. Subjects may be male or female. Women of childbearing potential must practice an acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, long-acting injectable contraceptive, double-barrier method (condom or intrauterine device [IUD] with spermicide), or partner's vasectomy.
6. Subjects must be between the ages of 18 and 55 years inclusive.
7. Subjects must be ambulatory, with a Kurtzke Expanded Disability Status Scale (EDSS) score between 0 and 5.0 inclusive.
8. Subjects must be willing and able to give written informed consent prior to entering the study.

Exclusion Criteria:

1. Long-term glatiramer acetate users who have been on therapy within 6 months of the baseline magnetic resonance imaging (MRI). New glatiramer acetate users who have initiated therapy for more than 6 weeks prior to the baseline MRI.
2. Previous use of cladribine.
3. Previous use of mitoxantrone.
4. Use of digitalis at study entry.
5. Previous use of immunosuppressive agents (such as azathioprine, cyclophosphamide or mycophenolate mofetil) in the last 6 months prior to screening.
6. Use of experimental or investigational drugs, including intravenous (IV) immunoglobulin within 6 months prior to screening.
7. Use of interferon agents within 1 month prior to the baseline MRI.
8. Use of corticosteroids (IV, intramuscular [IM] and/or by mouth [PO]) within 30 days prior to the baseline MRI.
9. Chronic corticosteroid (IV, IM and/or PO) treatment (more than 30 consecutive days) in the 6 months prior to the screening visit.
10. Subjects with diabetes.
11. Previous total body irradiation or total lymphoid irradiation.
12. Pregnancy or breast feeding.
13. Significant medical or psychiatric condition that affects the subject's ability to give informed consent, or to complete the study, or any condition which the investigator feels may interfere with participation in the study (e.g. alcohol or drug abuse).
14. Other diseases that can cause brain atrophy (ex. neurodegenerative disorder, cerebrovascular disease, history of alcohol abuse).
15. Bone density less than -2.5 standard deviations (SD) (osteoporosis).
16. A known history of sensitivity to mannitol.
17. Contraindication to, or known history of, sensitivity or severe reaction to steroids.
18. A known history of sensitivity to gadolinium.
19. Inability to successfully undergo MRI scanning.
20. Previous use of natalizumab.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 414 (Actual)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Stril, MD, Study Chair — Teva Neuroscience Canada

REFERENCES:
- [Result] Milo R, Panitch H. Combination therapy in multiple sclerosis. J Neuroimmunol. 2011 Feb;231(1-2):23-31. doi: 10.1016/j.jneuroim.2010.10.021. Epub 2010 Dec 15. PMID 21111490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GA + Placebo | GA + Prednisone
Started | 204 | 210
In Database as of January 29, 2009 | 199 | 209
Completed | 13 | 7
Not Completed | 191 | 203
Not completed — Ongoing: in database - January 29, 2009 | 131 | 109
Not completed — Ongoing: not in database - Jan 29, 2009 | 5 | 1
Not completed — Withdrawal by Subject | 13 | 47
Not completed — Teva requested participant withdrawal | 1 | 1
Not completed — Physician Decision | 8 | 7
Not completed — Non-compliance | 4 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 11 | 5
Not completed — Adverse Event | 8 | 18
Not completed — Death | 1 | 2
Not completed — Pregnancy | 3 | 0
Not completed — Other | 5 | 5

BASELINE CHARACTERISTICS:
Population: Represents database as of January 29, 2009
Groups:
- Total: Total of all reporting groups
Arm/Group | GA + Placebo | GA + Prednisone | Total
Number analyzed (Participants) | 199 | 209 | 408
Age, Customized [Number; unit: participants]
  <=29 years | 32 | 40 | 72
  =30 and < 40 years | 61 | 68 | 129
  =40 and < 50 years | 70 | 70 | 140
  =50 and < 55 years | 35 | 29 | 64
  >= 55 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 157 | 308
  Male | 48 | 52 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 10 | 9 | 19
  Asian / Oriental | 1 | 0 | 1
  Black of African Heritage | 13 | 15 | 28
  Caucasian | 171 | 179 | 350
  Other | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 1 | 5
  Canada | 16 | 20 | 36
  United States | 179 | 188 | 367
Time from First Multiple Sclerosis (MS) Symptom [Mean (Standard Deviation); unit: months] | 89.8 (104.5) | 76.7 (75.5) | 83.1 (91.0)
Time from MS Diagnosis [Mean (Standard Deviation); unit: months] | 40.5 (71.4) | 42.1 (62.9) | 41.3 (67.1)
T1 Enhancing Lesions at Baseline [Mean (Standard Deviation); unit: lesions] — Enhancing lesions represent new lesions due to recent disease activity and may indicate a relapse.
  171 GA + Placebo and 155 GA + Prednisone participants had baseline MRI data in the database as of January 29, 2009.
  lesions | 1.05 (2.77) | 1.86 (9.91) | 1.43 (7.12)
T1 Hypointense Lesions Volume at Baseline [Mean (Standard Deviation); unit: cm^3] — Hypointense lesions display as dark areas on the MRI image, and represent areas of permanent axonal damage.
  171 GA + Placebo and 155 GA + Prednisone participants had baseline MRI data in the database as of January 29, 2009.
  cm^3 | 0.94 (1.77) | 0.84 (1.50) | 0.89 (1.64)
T2 Lesions Volume at Baseline [Mean (Standard Deviation); unit: cm^3] — T2 lesions are hyperintense lesions meaning that they appear as bright spots on the MRI image. These tend to show the total number of lesions and disease burden.
  171 GA + Placebo and 155 GA + Prednisone participants had baseline MRI data in the database as of January 29, 2009.
  cm^3 | 5.51 (7.17) | 5.35 (7.97) | 5.44 (7.55)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Termination in Normalized Brain Volume Measured According to the SIENA (Structural Imaging Evaluation Using Normalization of Atrophy) Method
Description: Results represent the database as of January 29, 2009. Brain volume was measured at baseline and at months 24, 36 and at early termination visits by magnetic resonance imaging (MRI). Brain atrophy was measured by comparing the change in brain volume from baseline to the latest scan at the three during study timeframes. SIENA is a fully automated method of analyzing longitudinal brain change.
  Adjusted (least square) mean values are presented.
Time Frame: Day 0, latest scan at month 24, 36 or early termination visit
Population: Treated population of participants who had both a baseline MRI and an MRI at least one of the three during study time frames. The latest MRI was used if more than one during study MRI was available.
Measure: Least Squares Mean (Standard Error); unit: percent change of baseline brain volume
Arm/Group | GA + Placebo | GA + Prednisone
Number analyzed (Participants) | 105 | 84
percent change of baseline brain volume | -0.46 (0.088) | -0.43 (0.106)
Statistical Analysis 1: Comparison: GA + Placebo vs GA + Prednisone; Test type: Superiority or Other; p = 0.8023, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.26 to 0.20], Standard Error of Mean 0.11820976

2. Secondary Outcome: Cumulative Number of Enhancing Lesions at Months 12, 24 and 36
Description: Results represent the database as of January 29, 2009.
  Enhancing lesions are lesions that show inflammation on an MRI and are assumed to be new lesions. The sum of enhancing lesions observed in MRIs taken at months 12, 24 and 36 are offered.
Time Frame: Months 12, 24, and 36
Population: Treated population who had at least a 12 month MRI
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | GA + Placebo | GA + Prednisone
Number analyzed (Participants) | 155 | 143
lesions | 0.69 (3.28) | 0.76 (1.86)

3. Secondary Outcome: Change From Baseline to Month 36 or Early Termination Visit in Volume of T2-Lesions
Description: Results represent the database as of January 29, 2009.
  The difference in T2 brain lesion volume as observed in MRIs from baseline to Month 36 or the early termination visit. T2 lesions are hyperintense lesions meaning that they appear as bright spots on the MRI image. These tend to show the total number of lesions and disease burden.
Time Frame: Day 0, Month 36 or the early termination visit
Population: Treated population of participants with an MRI at the stated time frames.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | GA + Placebo | GA + Prednisone
Number analyzed (Participants) | 58 | 51
cm^3 | 0.07 (3.21) | 0.09 (2.93)

4. Secondary Outcome: Change From Baseline to Month 36 or Early Termination Visit in Volume of Hypointense Lesions
Description: Results represent the database as of January 29, 2009.
  The difference in hypointense brain lesion volume as observed in MRIs from baseline to Month 36 or the early termination visit. Hypointense lesions display as dark areas on the MRI image, and represent areas of permanent axonal damage.
Time Frame: Day 0, Month 36 or early termination visit
Population: Treated population of participants with an MRI at the stated time frames.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | GA + Placebo | GA + Prednisone
Number analyzed (Participants) | 58 | 51
cm^3 | 0.43 (1.60) | 0.17 (0.86)

ADVERSE EVENTS:
Time Frame: Day 1 through month 36
Arm/Group | GA + Placebo | GA + Prednisone
Serious Adverse Events (participants affected / at risk) | 16/199 | 13/209
Other Adverse Events (participants affected / at risk) | 131/199 | 151/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GA + Placebo (N=199) | GA + Prednisone (N=209)
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Closed head injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Multiple sclerosis (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GA + Placebo (N=199) | GA + Prednisone (N=209)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 5
Tachycardia (Cardiac disorders) | 0 | 6
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Colour blindness (Congenital, familial and genetic disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Tinnitis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Dry eye (Eye disorders) | 2 | 1
Lacrimation increased (Eye disorders) | 1 | 1
Madarosis (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 4
Eye allergy (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0
Asthenopia (Eye disorders) | 1 | 0
Optic atrophy (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Pupillary reflex impaired (Eye disorders) | 0 | 1
Macular cyst (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 9
Visual disturbance (Eye disorders) | 0 | 3
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 3
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 14
Dyspepsia (Gastrointestinal disorders) | 5 | 16
Epigastic discomfort (Gastrointestinal disorders) | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 7
Constipation (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 6
Enteritis (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Breath odour (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 15 | 15
Vomiting (Gastrointestinal disorders) | 6 | 7
Haematochezia (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0
Peritoneal lesion (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Administration site reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 13 | 21
Malaise (General disorders) | 0 | 6
Chills (General disorders) | 1 | 5
Peripheral coldness (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 5
Gait disturbance (General disorders) | 0 | 2
Chest discomfort (General disorders) | 3 | 5
Energy increased (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Feeling jittery (General disorders) | 1 | 3
Flushing (General disorders) | 1 | 1
Hangover (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 3
Irritability (General disorders) | 0 | 2
Swelling (General disorders) | 0 | 2
Thirst (General disorders) | 0 | 1
Inflammation (General disorders) | 2 | 0
Infusion site reaction (General disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 3
Injection site erythema (General disorders) | 9 | 3
Injection site haemorrhage (General disorders) | 0 | 1
Injection site induration (General disorders) | 3 | 1
Injection site mass (General disorders) | 1 | 0
Injection site nodule (General disorders) | 1 | 0
Injection site pain (General disorders) | 3 | 6
Injection site pruritus (General disorders) | 5 | 3
Injection site reaction (General disorders) | 8 | 8
Injection site swelling (General disorders) | 2 | 0
Injection site urticaria (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 4
Generalised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 3 | 5
Chest pain (General disorders) | 0 | 5
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 2 | 12
Adverse drug reaction (General disorders) | 1 | 2
Idiosyncratic drug reaction (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Allergy to animal (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 3
Food allergy (Immune system disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 3
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Vaginitis bacterial (Infections and infestations) | 2 | 0
Candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 2 | 3
Coxsackie viral infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 3 | 3
Tooth infection (Infections and infestations) | 2 | 2
Ear infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Conjunctivitis infective (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 4 | 2
Vaginal infection (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 2 | 3
Onychomycosis (Infections and infestations) | 2 | 0
Oral fungal infection (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 4
Herpes simplex (Infections and infestations) | 3 | 2
Herpes simplex ophthalmic (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 5 | 6
Bronchitis (Infections and infestations) | 13 | 5
Bronchitis acute (Infections and infestations) | 1 | 2
Bronchitis chronic (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0
Eczema infected (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 4
Pharyngitis streptococcal (Infections and infestations) | 2 | 1
Tinea infection (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 19 | 22
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 10 | 16
Upper respiratory tract infection (Infections and infestations) | 12 | 25
Cystitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 15 | 23
Bronchitis viral (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 3 | 3
Viral pharyngitis (Infections and infestations) | 0 | 2
Viral sinusitis (Infections and infestations) | 0 | 1
Caustic injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Injection site reaction (Injury, poisoning and procedural complications) | 1 | 0
Injection site urticaria (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 5
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 7
Accidental needle stick (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 2
Cardiac murmur (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 4 | 3
Heart rate decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Urine ketone body present (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Body temperature fluctuations (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 3 | 7
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 2
Protein total increased (Investigations) | 1 | 0
Blood testosterone decreased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1
Protein urine (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 0 | 1
Herpes simplex serology positive (Investigations) | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Increased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 6
Oedema (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 9
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 11
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Breast cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 4
Coordination abnormal (Nervous system disorders) | 0 | 2
Nystagmus (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 2
Circadian rhythm sleep disorder (Nervous system disorders) | 1 | 0
Hyperkinesia (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 14 | 31
Sinus headache (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 6
Migraine (Nervous system disorders) | 6 | 2
Multiple sclerosis (Nervous system disorders) | 2 | 0
Hypertonia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 11 | 12
Myoclonus (Nervous system disorders) | 2 | 0
Muscle spasticity (Nervous system disorders) | 4 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 7
Hypoaesthesia oral (Nervous system disorders) | 0 | 1
Lhermitte's sign (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 6 | 9
Diplegia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 6
Loss of proprioception (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 3 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 5 | 6
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 2 | 4
Agitation (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 4 | 9
Nervousness (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Tension (Psychiatric disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 10 | 9
Insomnia (Psychiatric disorders) | 22 | 44
Anger (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 3
Mood swings (Psychiatric disorders) | 1 | 3
Restlessness (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 2 | 2
Panic disorder (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 2
Abnormal dreams (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 2
Illusion (Psychiatric disorders) | 0 | 1
Claustrophobia (Psychiatric disorders) | 1 | 0
Speech disorder (Psychiatric disorders) | 0 | 1
Bruxism (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 6
Stress incontinence (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Hot flush (Reproductive system and breast disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 2
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine mass (Reproductive system and breast disorders) | 0 | 1
Genital pruritus female (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Laryngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 1
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Lipoatrophy (Skin and subcutaneous tissue disorders) | 3 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 12
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Alcohol use (Social circumstances) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 2 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Thyroid operation (Surgical and medical procedures) | 1 | 0
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 1
Uterine prolapse repair (Surgical and medical procedures) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 15
Hot flush (Vascular disorders) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 5
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.